CLINICAL TRIAL: NCT03037203
Title: A 4-Week, Double-blind, Placebo-controlled, Randomized, Multicenter, Crossover Study of the Safety, Efficacy, and Pharmacokinetics of JZP-110 [(R)-2-amino-3-phenylpropylcarbamate Hydrochloride] in Subjects With Parkinson's Disease and Excessive Sleepiness
Brief Title: A 4-Week Study of the Safety, Efficacy, and Pharmacokinetics of JZP-110 [(R)-2-amino-3-phenylpropylcarbamate Hydrochloride] in Subjects With Parkinson's Disease and Excessive Sleepiness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: JZP166-201
Record Dates: First submitted 2017-01-23; First posted 2017-01-31 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Excessive Sleepiness; Parkinson Disease
MeSH Terms: conditions — Disorders of Excessive Somnolence; Parkinson Disease | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): JZP-110 and Placebo
  Interventions: Drug: JZP-110; Other: Placebo
- Arm B (Experimental): JZP-110 and Placebo
  Interventions: Drug: JZP-110; Other: Placebo
- Arm C (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JZP-110 — 75 mg, 150 mg, 300 mg
  Arms: Arm A; Arm B
Other: Placebo

SUMMARY:
This study is a 4-week, multicenter, randomized, double-blind, placebo-controlled, ascending dose, 4-period crossover study designed to evaluate the safety, tolerability, efficacy, and PK of JZP-110 (75, 150, and 300 mg) in the treatment of excessive sleepiness in adult subjects with idiopathic PD.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic PD according to the UK PDS Brain Bank Criteria.
2. Hoehn and Yahr stage 1, 2, or 3.
3. Screening and Baseline ESS scores >11.

Exclusion Criteria:

1. Diagnosis of other degenerative Parkinsonian syndromes (e.g., progressive supranuclear palsy, multiple system atrophy [MSA], or dementia with Lewy bodies [DLB]).
2. Usual nightly time in bed of <6 hours, including the night before the Baseline visit.
3. Untreated or inadequately treated moderate to severe OSA.
4. Has evidence at screening of severe cognitive impairment or has cognitive impairment that in the opinion of the investigator would prevent completion of study procedures or the ability to provide informed consent.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-01; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Millie Gottwald, PharmD, Study Director — Jazz Pharmaceuticals
Locations (25):
- United States (25):
  - Southern California Institute For Respiratory Diseases, Inc., Los Angeles, California
  - Pacific Research Network, Inc, San Diego, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Rocky Mountain Movement Disorders Center, PC, Englewood, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - PAB Clinical Research, Brandon, Florida
  - MD Clinical, Hallandale, Florida
  - QPS MRA (Miami Research Associates), Miami, Florida
  - Bioclinica Research, Orlando, Florida
  - USF Health Byrd Institute, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Center for Sleep & Wake Disorders, Chevy Chase, Maryland
  - QUEST Research Institute, Farmington Hills, Michigan
  - Clinical Neurophysiology Services, P.C., Sterling Heights, Michigan
  - Henry Ford Medical Center - West Bloomfield, West Bloomfield, Michigan
  - St. Lukes Hospital Medical Center, Chesterfield, Missouri
  - Strong Sleep Disorders Center, Rochester, New York
  - Montefiore Sleep-Wake Disorders Center, The Bronx, New York
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Parkinson's Disease Research Unit - Thomas Jefferson University, Philadelphia, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina
  - Villages at Vanderbilt, Nashville, Tennessee
  - Evergreen Hospital Medical Center, Kirkland, Washington
  - Premier Clinical Research - Sherman, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Videnovic A, Amara AW, Comella C, Schweitzer PK, Emsellem H, Liu K, Sterkel AL, Gottwald MD, Steinerman JR, Jochelson P, Zomorodi K, Hauser RA. Solriamfetol for Excessive Daytime Sleepiness in Parkinson's Disease: Phase 2 Proof-of-Concept Trial. Mov Disord. 2021 Oct;36(10):2408-2412. doi: 10.1002/mds.28702. Epub 2021 Jun 30. PMID 34191352

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Sequence A: Subjects in Treatment Sequence A were assigned the following from Period 1, Week 1 through Period 4, Week 4: Placebo, JZP-110 75 mg, JZP 110 150 mg, and JZP 110 300 mg.
- Treatment Sequence B: Subjects in Treatment Sequence B were assigned the following from Period 1, Week 1 through Period 4, Week 4: JZP-110 75 mg, JZP 110 150 mg, JZP 110 300 mg, and Placebo.
- Treatment Sequence C: Subjects in Treatment Sequence C were assigned Placebo for each Period.
Period: Overall Study
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C
Started | 28 | 28 | 10
Completed | 27 | 26 | 9
Not Completed | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence A | Treatment Sequence B | Treatment Sequence C | Total
Number analyzed (Participants) | 28 | 28 | 10 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (7.64) | 62.9 (8.75) | 65.4 (9.75) | 64.6 (8.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 5 | 21
  Male | 18 | 22 | 5 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 1 | 4
  White | 27 | 24 | 9 | 60
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Early Discontinuation
Time Frame: Up to Day 35
Population: The Safety population includes all subjects who received at least one dose of study drug
Measure: Count of Participants; unit: Participants
Groups:
- JZP-110 75mg: The JZP-110 75 mg group consists of all subjects in the Safety population who also received at least 1 dose of 75 mg from Sequences A (28) and B (28), with a total of 56 subjects.
- JZP-110 150mg: The JZP-110 150 mg group consists of all subjects in the Safety population who also received at least 1 dose of 150 mg from Sequences A (28) and B (27), with a total of 55 subjects.
- JZP-110 300mg: The JZP-110 300 mg group consists of all subjects in the Safety population who also received at least 1 dose of 300 mg from Sequences A (28) and B (26), with a total of 54 subjects.
- Placebo: The Placebo group consists of all subjects in the Safety population who also received at least 1 dose of Placebo from Sequences A (28), B (26), and C (10) with a total of 64 subjects.
Arm/Group | JZP-110 75mg | JZP-110 150mg | JZP-110 300mg | Placebo
Number analyzed (Participants) | 56 | 55 | 54 | 64
Participants | 1 | 2 | 0 | 0

2. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score
Description: Change from Baseline ESS defined in terms of change from study baseline (prior to first dose in Period 1) to the end of each Treatment Period (Weeks 1, 2, 3, and 4).
  The Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions, asking subjects how likely they would be to doze off or fall asleep in different situations. Responses range from 0 = would never doze to 3 = high chance of dozing. Higher scores represent greater severity of excessive sleepiness. The total score ranges from 0 - 24, with higher scores representing greater severity of excessive sleepiness.
Time Frame: Baseline to Weeks 1, 2, 3, and 4
Population: The modified Intent-to-Treat population is defined as all randomized subjects who took at least one dose of study drug and have a Baseline and at least one post-Baseline efficacy assessment. Two subjects who did not have at least one post-baseline efficacy data were excluded from the mITT Population, resulting in a total of 64 subjects.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- JZP-110 75mg: The JZP-110 75 mg group consisted of all subjects in the mITT population from Sequences A (28 subjects) and B (27 subjects), for a total of 55 subjects.
- JZP-110 150mg: The JZP-110 150 mg group consisted of all subjects in the mITT population from Sequences A (28 subjects) and B (27 subjects), for a total of 55 subjects.
- JZP-110 300mg: The JZP-110 300 mg group consisted of all subjects in the mITT population from Sequences A (28 subjects) and B (27 subjects), for a total of 55 subjects.
- Placebo: The Placebo group includes all subjects in the mITT population from Sequences A, B, and C - 64 subjects in total.
Arm/Group | JZP-110 75mg | JZP-110 150mg | JZP-110 300mg | Placebo
Number analyzed (Participants) | 55 | 55 | 55 | 64
score on a scale | -4.82 (0.67) | -5.04 (0.70) | -5.72 (0.68) | -4.78 (0.58)

3. Other Pre Specified Outcome: Change From Baseline in the Mean Sleep Latency Time (in Minutes) on the Maintenance of Wakefulness Test (MWT)
Description: Change from Baseline mean sleep latency (in minutes) on the MWT defined in terms of change from study baseline (prior to first dose in Period 1) to the end of each Treatment Period (Weeks 1, 2, 3, and 4).
  The MWT is the standard objective measure of an individual's ability to remain awake during the daytime in a darkened, quiet environment. MWT sleep latency ranges from 0 to 40 minutes, with higher scores indicated greater ability to stay awake.
Time Frame: Baseline to Weeks 1, 2, 3, and 4
Population: The MWT analysis evaluated results from subjects in the mITT population who were in Group 1 only (N=53 subjects).
Measure: Least Squares Mean (Standard Error); unit: minutes
Groups:
- JZP-110 75mg: The JZP-110 75 mg group consisted of all subjects in the mITT population in Group 1 from Sequences A (24 subjects) and B (23 subjects), with a total of 47 subjects.
- JZP-110 150mg: The JZP-110 150 mg group consisted of all subjects in the mITT population in Group 1 from Sequences A (24 subjects) and B (23 subjects), with a total of 47 subjects.
- JZP-110 300mg: The JZP-110 300 mg group consisted of all subjects in the mITT population in Group 1 from Sequences A (24 subjects) and B (23 subjects), with a total of 47 subjects.
- Placebo: The Placebo group includes all subjects in the mITT population in Group 1 from Sequences A, B, and C - 53 subjects in total.
Arm/Group | JZP-110 75mg | JZP-110 150mg | JZP-110 300mg | Placebo
Number analyzed (Participants) | 47 | 47 | 47 | 53
minutes | 0.4289 (2.1254) | 2.6721 (2.1961) | 6.8133 (2.1351) | 1.7670 (1.8479)

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: The Safety population includes all subjects who received at least one dose of study drug
Groups:
- JZP-110 75 mg: The JZP-110 75 mg group consists of all subjects in the Safety population who also received at least 1 dose of 75 mg from Sequences A (28) and B (28), with a total of 56 subjects.
- JZP-110 150 mg: The JZP-110 150 mg group consists of all subjects in the Safety population who also received at least 1 dose of 150 mg from Sequences A (28) and B (27), with a total of 55 subjects.
- JZP-110 300 mg: The JZP-110 300 mg group consists of all subjects in the Safety population who also received at least 1 dose of 300 mg from Sequences A (28) and B (26), with a total of 54 subjects.
Arm/Group | JZP-110 75 mg | JZP-110 150 mg | JZP-110 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/55 | 0/54 | 0/64
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/55 | 1/54 | 0/64
Other Adverse Events (participants affected / at risk) | 4/56 | 5/55 | 4/54 | 0/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-110 75 mg (N=56) | JZP-110 150 mg (N=55) | JZP-110 300 mg (N=54) | Placebo (N=64)
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JZP-110 75 mg (N=56) | JZP-110 150 mg (N=55) | JZP-110 300 mg (N=54) | Placebo (N=64)
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 0
Dizziness (Nervous system disorders) | 3 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review trial results communications prior to public release and can embargo such communications for a period of at least 60 days from the time submitted to sponsor for review. If requested by sponsor, the PI will withhold publication for up to an additional 30 days. Furthermore, the first publication of study results must be a joint publication of all study sites unless a joint manuscript has not been submitted for publication within 12 months of completion of the study.

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT03037203/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03037203/SAP_001.pdf